CLINICAL TRIAL: NCT05793476
Title: Therapeutic Efficacy of Erbium:YAG Laser in Postpartum Patients With Episiotomy Scars in Respect of Genital Pelvic Pain and Scar Tissue Healing: A Randomized Sham-Controlled Prospective Study
Brief Title: Therapeutic Efficacy of Erbium:YAG Laser in Postpartum Patients With Episiotomy Scars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to find enough participants
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Principal Investigator, Cemal Tamer Erel, Clinical Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-83045809-604.01.01-416311
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Episiotomy Wound; Laser; Vulvodynia; Vulva Pain
Keywords: Episiotomy; Complications; Er-YAG Laser; Vulvodynia; Vulva Pain
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant doesn't know if she receives the sham or laser therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fotona Dynamis Er:YAG Laser System Arm (Experimental): Non-ablative thermal-only Er:YAG laser treatment using R11 and PS03 handpieces
  Interventions: Device: Fotona Dynamis Er:YAG Laser System
- Fotona Dynamis Er:YAG Laser System with Sham handpience (Sham Comparator): The same procedure is applied but with a sham handpiece.
  Interventions: Device: Fotona Dynamis Er:YAG Laser System with Sham handpiece

INTERVENTIONS:
Device: Fotona Dynamis Er:YAG Laser System — The patient receives 2940 nm Er:YAG Laser (XS Dynamis, Fotona, Slovenia) at intervals of 15-21 days. She receives 3 sessions, in total. 5% Lidocaine cream is applied 30 minutes before each procedure. Each session consists of application of R11 handpiece to the episiotomy scar at Turbo3 Micro Short Pulse mode, with spot size of 2 mm, fluence of 9.5-10 j/cm2, frequency of 2 Hz and 4 pulses per point and 3 passes followed by PS03 handpiece at Basic Long Pulse mode, with spot size of 5 mm, energy of 800 mJ, frequency of 1.4 Hz and 4 pulses per point and 2 passes.
  Arms: Fotona Dynamis Er:YAG Laser System Arm
Device: Fotona Dynamis Er:YAG Laser System with Sham handpiece — The same procedure is applied above but with a sham handpiece and parameter presentations masked.
  Arms: Fotona Dynamis Er:YAG Laser System with Sham handpience

SUMMARY:
Episiotomy is a planned surgical incision to the perineum and posterior wall of the vagina during the second stage of labor. The fibrotic and sclerotic scar tissue formed as part of the healing process of episiotomies may cause pain. Therefore, episiotomy is associated with sexual dysfunction due to the painful sexual intercourse, chronic pain and infections and scarring in long term. Er:YAG laser is a safe option for the treatment of vulvar pain.

Er:YAG laser is a non-invasive and non-ablative procedure that strengthens the connective tissue in the vaginal wall. It provides controlled thermal energy and causes shrinkage of collagen fibrils of the vaginal epithelium and lamina propria. It also induces neocollagenesis, elastogenesis and neoangiogenesis by temperature change. Er:YAG laser is also an effective modality to treat the scar tissue formed after the mediolateral episiotomy since it is a matter of functionality and esthetics. By tissue remodeling effect Er:YAG laser will improve the scar tissue of episiotomy and ameliorate the vulvar pain.

In this study, the therapeutic effect of Er:YAG laser on the tissue healing of the episiotomy scars and the reduction of vulvar pain.

DETAILED DESCRIPTION:
Episiotomy is a planned surgical incision to the perineum and posterior wall of the vagina during the second stage of labor. The fibrotic and sclerotic scar tissue formed as part of the healing process of episiotomies may cause pain. Therefore, episiotomy is associated with sexual dysfunction due to the painful sexual intercourse, chronic pain and infections and scarring in long term. 40% of the patients complain about persisted dyspareunia after 6 months of delivery. Genital pelvic pain/penetration disorders disturb the quality of sexual life of the couple and affect the psychology and wellbeing of the partners. Since, vulva is rich in afferent nerve endings, episiotomy scar healing is associated with pain. Er:YAG laser is a safe option for the treatment of vulvar pain.

Er:YAG laser is a non-invasive and non-ablative procedure that strengthens the connective tissue in the vaginal wall. It provides controlled thermal energy and causes shrinkage of the collagen fibrils in the vaginal epithelium and lamina propria. It also induces neocollagenesis, elastogenesis and neoangiogenesis by temperature change. With minimum damage to the peripheral tissue, the viable cells in the target tissue react to this temperature change by expressing heat shock proteins (HSP). Then, HSP increases the levels of transforming growth factor-beta, fibroblast growth factor, epidermal growth factor, platelet-derived growth factor, vascular epithelial growth factor which induce neocollagenesis and neoangiogenesis. Therefore, the thermal energy stored in the vaginal wall induces proliferation of the epithelium which is rich in glycogen, neovascularization and collagen production in the lamina propria. Er:YAG laser is also an effective modality to treat the scar tissue formed after the mediolateral episiotomy since it is a matter of functionality and esthetics. By tissue remodeling effect Er:YAG laser will improve the scar tissue of episiotomy and ameliorate the vulvar pain.

In this study, the therapeutic effect of Er:YAG laser on the tissue healing of the episiotomy scars and the reduction of vulvar pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult Female, 18 years of age or older
* Have given birth in the last 6 months with episiotomy
* Have vulvar pain and dyspareunia

Exclusion Criteria:

* History of connective tissue disease
* History of other diseases that can cause vulvar pain (neurological, dermatological, Infectious etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: Rate of change of pain | 6 months
  Change of vulvar pain in patients with mediolateral episiotomy measured by visual analogue scale (0-10)
Efficacy: Rate of scar tissue healing | 6 months
  Evaluation of the efficacy and safety of scar tissue healing by USG Elastography for fibrosis

SECONDARY OUTCOMES:
Efficacy: Rate of improvement in sexual function | 6 months
  Evaluation of the change of Genital Pelvic Pain by Female Sexual Function Index
Safety: Incidence and severity of device related Adverse Events | 6 months
  Incidence and severity of device related Adverse Events (i.e., infections, edema, superficial burns, wound dehiscence)

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Tamer Erel, Prof., Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No